CLINICAL TRIAL: NCT02720692
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, Multicenter, Evaluation of the Safety of N1539 Following Major Surgery
Brief Title: Evaluation of N1539 Following Major Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Baudax Bio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REC-15-017
Record Dates: First submitted 2016-03-22; First posted 2016-03-28 (Estimated); Results first posted 2023-05-25 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-05

CONDITIONS: Pain, Post-operative
Keywords: Pain; Analgesia; N1539; Phase 3
MeSH Terms: conditions — Pain, Postoperative; Pain; Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- N1539 30mg (Experimental): N1539 (Intravenous meloxicam) 30mg every 24 hours for up to 7 doses.
  Interventions: Drug: N1539
- IV Placebo (Placebo Comparator): IV Placebo every 24 hours for up to 7 doses.
  Interventions: Drug: Intravenous Placebo

INTERVENTIONS:
Drug: N1539
  Other Names: Intravenous meloxicam
  Arms: N1539 30mg
Drug: Intravenous Placebo
  Arms: IV Placebo

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of N1539 in a variety of post-surgical conditions.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily provide written informed consent.
* Male or female between 18 and 80 years of age, inclusive.
* Be planning to undergo major elective surgery, and be expected to require intravenous analgesia and remain in an inpatient setting for at least 24-48 hours and are expected to receive at least two study doses.
* Female subjects are eligible only if all the following apply:

  * Not pregnant;
  * Not breastfeeding;
  * Not able to become pregnant;
  * Not planning to become pregnant during the study or 28 day follow up;
  * Commit to the use of an acceptable form of birth control for the duration of the study.
* Have a body mass index ≤40 kg/m2
* Be able to understand the study procedures, comply with all study procedures, and agree to participate in the study program.
* For oncology cases, have a histologically confirmed diagnosis of a primary solid tumor, affecting any one of the following organs: breast, skin, colon, prostate, uterus, ovaries, urethra, penis, or vulva; AND based on clinical, laboratory, radiologic, pathologic, and surgical findings, the tumor is confined to the primary organ, without evidence of local, regional or distal spread; AND have a performance status such that they are able to carry on normal activities of daily life without limitations.

Exclusion Criteria:

* Have a known allergy to meloxicam or any excipient of N1539, aspirin, other non-steroidal anti-inflammatory drugs (NSAIDs).
* Be scheduled to undergo cranial surgery, open heart procedure, any type of coronary artery bypass graft, organ transplant, or any other surgical procedure in which NSAIDs are contraindicated.
* Planned or actual admission to the intensive care unit at any time during study participation.
* Have clinically significant laboratory abnormalities.
* Have a history of myocardial infarction within the preceding 12 months.
* Have history of HIV, or hepatitis B or C.
* Have a history or clinical manifestations of significant renal, hepatic, cardiovascular, metabolic, neurologic, psychiatric, respiratory, or other condition that would preclude participation in the study.
* Have active or recent (within 6 months) gastrointestinal ulceration or bleeding
* Have a known bleeding disorder which may be worsened with the administration of a NSAID.
* Have evidence of a clinically significant 12 lead ECG abnormality.
* Have a history of alcohol abuse (regularly drinks > 4 units of alcohol per day; 8 oz. beer, 3 oz. wine, 1 oz. spirits) or a history of prescription/illicit drug abuse within the past 5 years.
* Have positive results on the urine drug screen for cocaine or PCP or alcohol breath test indicative of illicit drug or alcohol abuse.
* Unable to discontinue medications, that have not been at a stable dose for at least 14 days prior to the scheduled surgical procedure, within 5 half-lives of the specific prior medication (or, if half-life is not known, within 48 hours) before dosing with study medication.
* Be unable to discontinue herbal medications at least 7 days prior to surgery through last dose of study medication.
* Be receiving lithium, or a combination of furosemide with either an angiotensin converting enzyme inhibitor or an angiotensin receptor blocker
* Be currently receiving treatment with oral meloxicam (Mobic®) or other NSAID within 7 days prior to surgery.
* Have received any investigational product within 30 days before dosing with study medication.
* Have previously received N1539 in clinical trials, or had major surgery in the last 3 months that would interfere with study assessments.
* Have undergone or be expected to undergo radiation therapy, chemotherapy, or other biological therapy for cancer treatment, within 60 days prior to screening, through the last study visit, approximately 30 days after dosing.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 722 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (30):
- United States (19):
  - Florence, Alabama
  - Montgomery, Alabama
  - Sheffield, Alabama
  - Gilbert, Arizona
  - Phoenix, Arizona
  - Anaheim, California
  - Bakersfield, California
  - Miami, Florida
  - Tamarac, Florida
  - Tampa, Florida
  - Chicago, Illinois
  - Great Falls, Montana
  - Cleveland, Ohio
  - Columbus, Ohio
  - Tyrone, Pennsylvania
  - Hendersonville, Tennessee
  - Houston, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
- Australia (4):
  - Chermside, Queensland
  - Kippa-Ring, Queensland
  - Southport, Queensland
  - Richmond, Victoria
- Canada (4):
  - Halifax, Nova Scotia
  - Kingston, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
- New Zealand (3):
  - Auckland
  - Christchurch
  - Hamilton

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sharpe KP, Berkowitz R, Tyndall WA, Boyer D, McCallum SW, Mack RJ, Du W. Safety, Tolerability, and Effect on Opioid Use of Meloxicam IV Following Orthopedic Surgery. J Pain Res. 2020 Jan 21;13:221-229. doi: 10.2147/JPR.S216219. eCollection 2020. PMID 32021411
- [Derived] Bergese SD, Melson TI, Candiotti KA, Ayad SS, Mack RJ, McCallum SW, Du W, Gomez A, Marcet JE. A Phase 3, Randomized, Placebo-Controlled Evaluation of the Safety of Intravenous Meloxicam Following Major Surgery. Clin Pharmacol Drug Dev. 2019 Nov;8(8):1062-1072. doi: 10.1002/cpdd.666. Epub 2019 Feb 20. PMID 30786162
- [Derived] Viscusi ER, Gan TJ, Bergese S, Singla N, Mack RJ, McCallum SW, Du W, Hobson S. Intravenous meloxicam for the treatment of moderate to severe acute pain: a pooled analysis of safety and opioid-reducing effects. Reg Anesth Pain Med. 2019 Mar;44(3):360-368. doi: 10.1136/rapm-2018-100184. Epub 2019 Feb 7. PMID 30737315

RESULTS

PARTICIPANT FLOW:
Groups:
- N1539 30 mg: N1539 (Intravenous meloxicam) 30 mg every 24 hours for up to 7 doses.
  N1539
- IV Placebo: IV Placebo every 24 hours for up to 7 doses.
  Intravenous Placebo
Period: Overall Study
Arm/Group | N1539 30 mg | IV Placebo
Started | 539 | 183
Treated | 538 | 183
Completed Treatment | 519 | 177
Completed | 526 | 180
Not Completed | 13 | 3
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Lost to Follow-up | 8 | 3
Not completed — Subject unable to return for visit | 1 | 0

BASELINE CHARACTERISTICS:
Population: All Treated Subjects (Safety Analysis Set)
Groups:
- Total: Total of all reporting groups
Arm/Group | N1539 30 mg | IV Placebo | Total
Number analyzed (Participants) | 538 | 183 | 721
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 0 | 2
  Between 18 and 65 years | 416 | 140 | 556
  >=65 years | 120 | 43 | 163
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.9 (13.56) | 53.0 (13.77) | 53.0 (13.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 315 | 113 | 428
  Male | 223 | 70 | 293
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 76 | 29 | 105
  Not Hispanic or Latino | 462 | 154 | 616
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 7 | 4 | 11
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 68 | 21 | 89
  White | 459 | 155 | 614
  More than one race | 1 | 3 | 4
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 502 | 168 | 670
  Canada | 5 | 3 | 8
  New Zealand | 8 | 2 | 10
  Australia | 23 | 10 | 33
Advanced Age (>65) with Impaired Renal Function (GFR<90) [Count of Participants; unit: Participants] | 88 | 31 | 119
Surgery Site/Type [Count of Participants; unit: Participants]
  Orthopedic | 273 | 93 | 366
  Abdominal/Pelvic | 254 | 87 | 341
  Spinal | 10 | 3 | 13
  Other | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Adverse Events
Description: Number of subjects reporting 1 or more treatment-emergent adverse events
Time Frame: 28 Days
Population: All Treated Subjects (Safety Analysis Set)
Measure: Count of Participants; unit: Participants
Arm/Group | N1539 30 mg | IV Placebo
Number analyzed (Participants) | 538 | 183
Participants | 339 | 119

2. Secondary Outcome: Investigator Satisfaction With Surgical Wound Healing
Description: Investigators assessed their satisfaction with the healing of the surgical wound according to an 11-point numeric rating scale (0-10) where a score of 0 was completely unsatisfied (worse outcome), and a score of 10 was completely satisfied (better outcome).
Time Frame: Up to 7 days after last study dose
Population: All Treated Subjects (Safety Analysis Set)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | N1539 30 mg | IV Placebo
Number analyzed (Participants) | 538 | 183
score on a scale
  One day after last study dose/Discharge | 9.5 (0.88) | 9.4 (0.97)
  7 Days after last study dose | 9.3 (1.18) | 9.4 (0.86)

3. Secondary Outcome: Postoperative Opioid Use
Description: Postoperative opioid use was measured throughout the inpatient phase and converted to the total IV morphine equivalent dose
Time Frame: Up to 7 days
Population: All Treated Subjects (Safety Analysis Set)
Measure: Mean (Standard Deviation); unit: mg (IV Morphine Equivalent Dose)
Arm/Group | N1539 30 mg | IV Placebo
Number analyzed (Participants) | 538 | 183
mg (IV Morphine Equivalent Dose)
  Day 1 (Hour 0-24) | 17.0 (22.10) | 21.8 (24.70)
  Day 2 (Hour 24-48) | 8.6 (19.15) | 11.3 (21.82)
  Day 3 (Hour 48-72) | 4.1 (16.60) | 6.2 (21.83)
  Day 1-2 (Hour 0-48) | 25.3 (36.96) | 32.7 (41.44)
  Day 1-3 (Hour 0-72) | 27.4 (44.67) | 35.9 (52.77)
  During Treatment | 28.8 (57.39) | 37.5 (66.06)
Statistical Analysis 1: Comparison: N1539 30 mg vs IV Placebo; Test type: Superiority; p < 0.05, ANCOVA — P<0.05 applies to Day 1 (0-24 Hours; p=0.0033), Days 1-2 (0-48 Hours; p=0.0077), and Days 1-3 (0-72 Hours; p=0.0152)

ADVERSE EVENTS:
Time Frame: AE data were collected from the time of first study dose, through the last study contact, 28 days following the last study dose.
Arm/Group | N1539 30 mg | IV Placebo
All-Cause Mortality (participants affected / at risk) | 0/538 | 0/183
Serious Adverse Events (participants affected / at risk) | 14/538 | 10/183
Other Adverse Events (participants affected / at risk) | 227/538 | 85/183
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | N1539 30 mg (N=538) | IV Placebo (N=183)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Jejunal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Omental infarction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0)
Hepatocellular injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Abdominal abscess (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Incision site infection (Infections and infestations) | 1 (1) | 0 (0)
Mesenteric abscess (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Postoperative abscess (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Anastomotic ulcer (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural pulmonary embolism (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Postoperative ileus (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Tendon injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 1 (1)
Hypervolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | N1539 30 mg (N=538) | IV Placebo (N=183)
Anaemia (Blood and lymphatic system disorders) | 18 (18) | 4 (4)
Constipation (Gastrointestinal disorders) | 51 (51) | 17 (17)
Vomiting (Gastrointestinal disorders) | 27 (30) | 14 (15)
Nausea (Gastrointestinal disorders) | 123 (129) | 50 (57)
Alanine aminotransferase increased (Investigations) | 11 (11) | 7 (7)
Gamma-glutamyltransferase increased (Investigations) | 21 (21) | 5 (5)
Dizziness (Nervous system disorders) | 15 (15) | 7 (8)
Headache (Nervous system disorders) | 20 (21) | 12 (13)
Insomnia (Psychiatric disorders) | 9 (9) | 6 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 21 (21) | 10 (10)
Hypotension (Vascular disorders) | 9 (9) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Discussion and/or publication of data generated is not permitted without the prior written consent of the sponsor.

DOCUMENTS (2):
  • Study Protocol (2016-07-13): https://cdn.clinicaltrials.gov/large-docs/92/NCT02720692/Prot_000.pdf
  • Statistical Analysis Plan (2017-02-17): https://cdn.clinicaltrials.gov/large-docs/92/NCT02720692/SAP_001.pdf